CLINICAL TRIAL: NCT02551354
Title: Estimation of Pain During Epidural Analgesia During Labor - a Monocentric Study
Brief Title: Estimation of Pain During Epidural Analgesia During Labor
Acronym: PERIDANS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1208078
Record Dates: First submitted 2015-09-11; First posted 2015-09-16 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2015-09

CONDITIONS: Labor, Obstetric; Pain
Keywords: Labor, Obstetric; pain; pupil diameter; Visual Analogic Scale (VAS)
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Pain assess by :
  * Visual Analogic Scale (VAS).
  * Portable video pupillometer
  Interventions: Device: Portable video pupillometer

INTERVENTIONS:
Device: Portable video pupillometer — Portable video pupillometer measures pupil diameter (PD) in patient during obstetrical labor

SUMMARY:
Epidural regional anesthesia is a technique to eliminate or lessen pain during obstetric labor and childbirth. It consists in establishing a catheter into the epidural space and to block the transmission of pain sensations by injecting a local anesthetic and an opioid. In 10-25% of cases the epidural does not give perfect results, causing it to test its effectiveness, which is mainly done by questioning the patient on mitigation or disappearance of pain. This collaboration of patients is sometimes limited in our care structure by the inability to assess or express the pain, mainly due to cultural differences or language barriers, which can represent up to 15% of women in our institution. This led to develop objective measures of pain techniques used at the bedside.

Pupil diameter (PD) varies under the double influence of sympathetic system (Σ), dilator of the pupil, and parasympathetic system (pΣ).

The PD increases in response to painful stimulation, in proportion to the intensity of the nociceptive stimulus. This variation of PD has been proposed as a means of evaluation of pain in patients under general anesthesia, but has been little studied in conscious subjects.

There are other permanent changes in the PD, due to constant interaction between Σ and pΣ systems. Few data have been published to date on this PD variability (PDV).

ELIGIBILITY:
Inclusion Criteria:

* Obstetrical Labor
* Able to rate their pain using VAS
* dilatation of the cervix under 6 centimeters
* Written consent

Exclusion Criteria:

* - Not having a anesthesia consultation during the 48 hours before delivery
* With a contra-indication for an epidural
* To which an incident occurred during a previous epidural using a medication used in the study
* Operated a unilateral or bilateral ocular surgery modifying the possibilities of variation of pupil diameter
* general anesthesia in the seven days preceding delivery
* Carry a pacemaker or heart grafted
* Having Parkinson's disease history, insulin or non-insulin diabetes or chronic alcoholism
* Having cardiac arrhythmia (atrial fibrillation or frequent extrasystoles)
* Treated for hypertension by receptor antagonists of angiotensin type 2
* anti-arrhythmic treatment or blocker,
* Refusing to participate in the study
* With a contra-indication for the use of ropivacaine and sufentanil.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Pupil diameter variability | From baseline to fifteen minutes after start of Epidural regional anesthesia
  Compare Pupil Diameter Variability (PDV) measured before Epidural regional anesthesia and after Epidural regional anesthesia. PDV is aera under the curve of Pupil Diameter from start of the contraction (baseline) to time to peak of the contraction.

SECONDARY OUTCOMES:
pupil diameter | From baseline to fifteen minutes after start of Epidural regional anesthesia
  Compare the Pupil Diameter measured five seconds after time to peak of contraction before Epidural regional anesthesia and after Epidural regional anesthesia
Visual Analogic Scale (VAS) | From baseline to fifteen minutes after start of Epidural regional anesthesia
  Compare the VAS measured at the end of contraction before Epidural regional anesthesia and after Epidural regional anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: David Charier, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France